CLINICAL TRIAL: NCT00939484
Title: A Phase II Clinical Trial Evaluating the Efficacy and Safety of GDC-0449 in Adults With Recurrent or Refractory Medulloblastoma
Brief Title: Vismodegib in Treating Patients With Recurrent or Refractory Medulloblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03020; NCI-2012-03020 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-025B (Other: Pediatric Brain Tumor Consortium); PBTC-025B (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-03

CONDITIONS: Adult Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — HhAntag691

ARMS (1):
- Treatment (vismodegib) (Experimental): Patients receive vismodegib PO once daily on days 1-28. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Pharmacological Study; Drug: Vismodegib

INTERVENTIONS:
Other: Pharmacological Study — Correlative studies
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This phase II trial is studying how well vismodegib works in treating adult patients with recurrent or refractory medulloblastoma. Vismodegib may slow the growth of tumor cells and may be an effective treatment for medulloblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the efficacy of GDC-0449 (vismodegib) treatment for adult patients with recurrent or refractory medulloblastoma, as measured by the objective response rates for patients without (Stratum A) and with (Stratum B) evidence of activation of Sonic Hedgehog (SHH) signaling pathway tumors.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of GDC-0449 administered on a once daily schedule.

II. To estimate the duration of objective response and progression-free survival (PFS).

III. To characterize the pharmacokinetics (plasma and cerebrospinal fluid) of GDC-0449 in adults with refractory medulloblastoma.

IV. To document pathologic and genomic methods to identify CNS tumors with activation of the PTCH/SHH pathway.

V. To describe the objective responses observed in patients whose pathologic assessment of tumor result in unknown (Stratum C) evidence of activation of Sonic Hedgehog (SHH) signaling pathway tumors.

OUTLINE: This is a multicenter study. Patients are stratified according to PTCH/Sonic Hedgehog signaling pathway activation (inactivated vs activated vs unknown).

Patients receive vismodegib orally (PO) once daily on days 1-28. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of medulloblastoma (including posterior fossa PNET) that is recurrent, progressive, or refractory to standard therapy and for which there is no known curative therapy are eligible; there must be evidence of residual measurable disease or lesion in pre-study MRI as described in section; patients with spinal disease that is measurable will be eligible
* The diagnosis should be confirmed at the treating institution and tissue (either from the diagnosis or relapse or preferably from both time points) must be available for biological studies
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration; this is to be documented in the database
* Eastern Cooperative Oncology Group (ECOG) performance status 0- 2
* No other myelosuppressive chemotherapy or immunotherapy within 4 weeks prior to study entry (6 weeks if prior nitrosourea)
* Decadron dose should also be stable or decreasing for at least 1 week (7days) prior to starting therapy
* Radiation therapy (XRT) >= 3 months prior to study entry for craniospinal irradiation (>= 23 Gy); >= 8 weeks for local irradiation to primary tumor; >= 2 weeks prior to study entry for focal irradiation for symptomatic metastatic sites
* Off all colony stimulating factors >= 1 week prior to study entry (GCSF, GM CSF, erythropoietin)
* Absolute neutrophil count (ANC) >= 1000/μL
* Platelet count >= 50,000/uL (transfusion independent)
* Hemoglobin >= 8.0 gm/dL (may receive RBC transfusions)
* Creatinine clearance or radio-isotope GFR >= 70ml/min/1.73 m2 or
* A serum creatinine =< 2.0 mg/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x institutional ULN
* Serum glutamic-oxalacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 times institutional ULN
* Serum albumin >= 2.5 g/dL
* Patient must have recovered from the significant acute toxicities of all prior therapy before entering this study and meet all other eligibility criteria
* Pregnancy should be avoided for 12 months after the last dose of GDC-0449 for females of child-bearing potential; female patients of childbearing potential must not be pregnant or breast-feeding; female patients of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to beginning treatment
* Women of childbearing potential are required to use 2 forms of acceptable contraception, including one barrier method during participation in the study and for the 12 months following the last dose; for medical or personal reasons, 100% commitment to abstinence is considered an acceptable form of birth control. All patients should receive contraceptive counseling either by the investigator, or by an OB/gynecologist or other physician who is qualified in this area of expertise; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the of GDC-0449 to cause spontaneous abortion or birth defects
* Signed informed consent according to institutional guidelines must be obtained

Exclusion Criteria:

* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results
* Patients receiving any other anticancer or investigational drug therapy
* Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy
* Life expectancy < 12 weeks as determined by treating physician
* Inability to swallow capsules
* Prior treatment with GDC-0449 or other antagonists of the HH pathway
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* History of congestive heart failure
* History of ventricular arrhythmia requiring medication
* Uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution despite adequate electrolyte supplementation
* Congenital long QT syndrome

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (13):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Pediatric Brain Tumor Consortium, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Robinson GW, Orr BA, Wu G, Gururangan S, Lin T, Qaddoumi I, Packer RJ, Goldman S, Prados MD, Desjardins A, Chintagumpala M, Takebe N, Kaste SC, Rusch M, Allen SJ, Onar-Thomas A, Stewart CF, Fouladi M, Boyett JM, Gilbertson RJ, Curran T, Ellison DW, Gajjar A. Vismodegib Exerts Targeted Efficacy Against Recurrent Sonic Hedgehog-Subgroup Medulloblastoma: Results From Phase II Pediatric Brain Tumor Consortium Studies PBTC-025B and PBTC-032. J Clin Oncol. 2015 Aug 20;33(24):2646-54. doi: 10.1200/JCO.2014.60.1591. Epub 2015 Jul 13. PMID 26169613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was distributed to the sites on June 18, 2009, and received the first IRB approval on July 20, 2009. The study was closed to accrual on December 07, 2012. Thirty two (32) patients have been enrolled to the study, Last patient went off treatment in October 2013.
Pre-assignment Details: Total 32 patients were registered on this study, 8 in Stratum A, 21 in Stratum B and 3 in Stratum C. One patient in Stratum B was declared ineligible.
Groups:
- Stratum A (PTCH/SHH Pathway Inactivated): Adult patients with recurrent or refractory medulloblastoma who have tumors without evidence of PTCH/SHH pathway activation
- Stratum B (PTCH/SHH Pathway Activated): Adult patients with recurrent or refractory medulloblastoma who have tumors with evidence of activation of the PTCH/SHH pathway
- Stratum C (Unknown PTCH/SHH Pathway Activation): Adult patients with recurrent or refractory medulloblastoma registered on protocol whose tumor assay is inconclusive as to whether or not the PTCH/SHH pathway is activated or whose tissue sample is inadequate to assess the PTCH/SHH pathway status
Period: Overall Study
Arm/Group | Stratum A (PTCH/SHH Pathway Inactivated) | Stratum B (PTCH/SHH Pathway Activated) | Stratum C (Unknown PTCH/SHH Pathway Activation)
Started | 8 | 20 | 3
Completed | 0 | 0 | 0
Not Completed | 8 | 20 | 3
Not completed — Progression/Relapse | 8 | 20 | 3

BASELINE CHARACTERISTICS:
Population: One patient in Stratum B was ineligible for the study and thus was not included in the baseline table.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum A (PTCH/SHH Pathway Inactivated) | Stratum B (PTCH/SHH Pathway Activated) | Stratum C (Unknown PTCH/SHH Pathway Activation) | Total
Number analyzed (Participants) | 8 | 20 | 3 | 31
Age, Continuous [Median (Full Range); unit: years] — Age at study enrollment
  years | 23.8 [22.4 to 40.6] | 32.0 [23.5 to 51.9] | 32.9 [25.3 to 38.6] | 30.3 [22.4 to 51.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 2 | 13
  Male | 6 | 11 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 18 | 2 | 27
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 3
  White | 7 | 16 | 3 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 20 | 3 | 31
Diagnosis [Number; unit: participants]
  Desmoplastic medulloblastoma | 0 | 1 | 0 | 1
  Medulloblastoma, NOS | 8 | 18 | 3 | 29
  Primitive neuroectodermal tumor | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (CR+PR) Sustained for ≥ 8 Weeks
Description: Objective response is either a complete response or a partial response sustained for 8 weeks in a patient. The objective response rate will be reported separately for patients of each stratum. CR is complete disappearance of all enhancing tumor. PR is >= 50% reduction in tumor size.
Time Frame: Up to 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Stratum A (PTCH/SHH Pathway Inactivated) | Stratum B (PTCH/SHH Pathway Activated) | Stratum C (Unknown PTCH/SHH Pathway Activation)
Number analyzed (Participants) | 8 | 20 | 3
proportion of participants | 0 [0 to 0.37] | 0.15 [0.03 to 0.38] | 0 [0 to 0.71]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is measured from the date of initial treatment with GDC-0449 until the earliest of progression or death on study. PFS is censored at the last tumor assessment date for patients without disease progression who have not died within 30 days of last exposure to study treatment. Kaplan-Meier method is used to estimate the progression-free survival.
Time Frame: From start of treatment up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum A (PTCH/SHH Pathway Inactivated) | Stratum B (PTCH/SHH Pathway Activated) | Stratum C (Unknown PTCH/SHH Pathway Activation)
Number analyzed (Participants) | 8 | 20 | 3
months | 1.64 [0.43 to 1.84] | 2.76 [1.38 to 6.38] | 1.48 [1.38 to 1.84]

3. Secondary Outcome: Duration of Objective Response
Description: The duration of objective response is measured from the initial scan documenting complete or partial response that was subsequently confirmed until the earlier of documented progression or death on study. Duration of objective response is censored at the last tumor assessment date for patients without disease progression who have not died within 30 days of last exposure to study treatment.
Time Frame: From start of treatment up to 2 years
Population: Patients with sustained objective response
Measure: Median (Full Range); unit: months
Arm/Group | Stratum B (PTCH/SHH Pathway Activated)
Number analyzed (Participants) | 3
months | 4.59 [1.48 to 4.77]

4. Secondary Outcome: Pharmacokinetic Parameters of Vismodegib, CSF Penetration
Description: The estimated median of cerebrospinal fluid (CSF) drug penetration is reported when expressed as an AUC ratio of CSF vismodegib to that of unbound drug in plasma.
Time Frame: up to 12 month
Population: The calculation of drug penetration is based on patients who had the course 1 plasma and CSF drug concentration data
Measure: Median (Full Range); unit: ratio
Groups:
- PBTC025B: Adult patients with a histologically confirmed diagnosis of medulloblastoma (including posterior fossa PNET) that is recurrent, progressive, or refractory.
Arm/Group | PBTC025B
Number analyzed (Participants) | 28
ratio | 0.12 [0.03 to 0.28]

ADVERSE EVENTS:
Time Frame: Adverse events were collected non-systematically for each of the participants from the time of enrollment to the completion of therapy or to the time off study.
Arm/Group | Stratum A (PTCH/SHH Pathway Inactivated) | Stratum B (PTCH/SHH Pathway Activated) | Stratum C (Unknown PTCH/SHH Pathway Activation)
Serious Adverse Events (participants affected / at risk) | 5/8 | 12/20 | 3/3
Other Adverse Events (participants affected / at risk) | 8/8 | 20/20 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A (PTCH/SHH Pathway Inactivated) (N=8) | Stratum B (PTCH/SHH Pathway Activated) (N=20) | Stratum C (Unknown PTCH/SHH Pathway Activation) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Death NOS (General disorders) | 1 (1) | 2 (2) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Hypoglossal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A (PTCH/SHH Pathway Inactivated) (N=8) | Stratum B (PTCH/SHH Pathway Activated) (N=20) | Stratum C (Unknown PTCH/SHH Pathway Activation) (N=3)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 4 (8) | 1 (2)
Cardiac disorders - Other, specify[Right Bundle Branch Block] (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eye disorders - Other, specify[Bilateral Proptosis] (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify[assymetric pupils and conjunctival injection] (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 7 (11) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (8) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 7 (12) | 3 (6)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 8 (12) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify[presssure back of head] (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 6 (8) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 11 (39) | 2 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 6 (13) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 7 (12) | 0 (0)
Weight loss (Investigations) | 0 (0) | 2 (4) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 9 (26) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 7 (10) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 7 (12) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 5 (6) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 5 (6) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5) | 6 (18) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify[right upper extremity weakness] (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 9 (10) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 10 (12) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (3) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Psychiatric disorders - Other, specify[nightmare one time] (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify[urinary hesitancy] (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less